CLINICAL TRIAL: NCT05059184
Title: Long-term Sequelae of COVID-19 (Myalgic Encephalomyelitis): An International Cross-Sectional Study
Acronym: ME
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Shaheen, Ahmed Shaheen, Alexandria University
Other Study IDs: KRL-HI-ERC/Sep21/03
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Myalgic Encephalomyelitis
Keywords: Long covid syndrome; Myalgic Encephalomyelitis; chronic fatigue syndrome; symptoms of COVID-19
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Methods

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This is an observational cross-sectional study, there is no need for intervention — This is an observational cross-sectional study. There is no need for intervention

SUMMARY:
The term recovery from COVID-19 caused by SARS-CoV-2 is unverified because the infection leaves many symptoms due to permanent effects on multiple organs; The primary objective of this research is to understand acute and chronic long COVID symptoms by asking questions detecting patient's experience especially symptoms lasting for several months which is known as chronic fatigue syndrome(Myalgic encephalitis). The study focuses on symptoms describing Myalgic encephalitis which may still affect COVID patients for several months after the infection along with making a big picture about rare symptoms that may the patient experienced during or after the infection.

A secondary objective of this research is to focus on the long-term sequelae effects and comorbidities following COVID-19 vaccination.

DETAILED DESCRIPTION:
After the appearance of COVID-19 caused by SARS-CoV-2, the pandemic has spread and had a profound effect on the lives and health of people around the Whole world causing around 3.97 million deaths and more than 183 million confirmed cases of the covid-19. The pandemic of COVID-19 may leave unexplainable symptoms after recovery. COVID-19 pandemic has a lot of serious symptoms, but some last for some time even after the recovery. Even some of the people who had mild symptoms during COVID-19 continue to have long terms effects after initial recovery. These people are called "long haulers" and these symptoms are called Long COVID-19. Long haulers still suffer from permanent symptoms due to multi-organ dysfunction despite normal nucleic acid tests that detect the virus.

According to Dr. Anthony Fauci "patients with COVID-19 can develop a post-viral syndrome that's very strikingly similar to Myalgic encephalomyelitis/chronic fatigue syndrome" Long COVID-19 involves multiple organs and affects many systems mainly respiratory, cardiovascular, neurological, gastrointestinal, and musculoskeletal systems. The symptoms of long-covid include shortness of breath, cough, myalgias, disturbances in the sense of taste and smell, fatigue, fever, chills, and, less commonly, rhinitis and gastrointestinal symptoms cardiac abnormalities, cognitive impairment, sleep disturbances, symptoms of post-traumatic stress disorder, muscle pain, concentration problems, and headache. Those manifestations persist in one of 10 patients of the infection and last for 3-4 weeks of acute symptoms and chronic symptoms last for more than 12 weeks after the infection. According to The Centers for Disease Control and Prevention (CDC), 150 patients out of 300 who were PCR-positive for SARS-CoV-2 had permanent symptoms after three weeks after the positive test.

In case the fatigue persists for six months, it is called Myalgic Encephalomyelitis / Chronic Fatigue Syndrome (ME/CFS).

Although the period of 6 months is no longer required for ME diagnosis according to 2011's ME international Consensus Criteria, it is still common in literature.

Chronic fatigue syndrome /post-viral myalgia can not only covid-19 but also follow viral infections such as Epstein-Barr virus, Ross River virus, enteroviruses, human herpesvirus, Ebola virus, West Nile virus, Dengue virus, and parvovirus; bacteria, such as Borrelia burgdorferi, Coxiella burnetii, and Mycoplasma pneumonia; and sometimes parasites, such as Giardia lamblia, so it is expected but the problem is that it is unknown how severe it is or how it can affect the public health.

Recently, there has been global concern about the effectiveness and safety of COVID-19 vaccines. According to WHO, the most common side effects that were reported about COVID-19 vaccines were fever, fatigue, headache, muscle pain, chills, diarrhea, and pain at the injection site which is more or less like some of the post covid infection symptoms so it was found that it is logical to add a section to gather information about the vaccine status, type, and timing with the symptoms.

Also, some cases were reported from Canada reported weird and rare symptoms like Beau lines.

ELIGIBILITY:
Inclusion Criteria:

* • Persons had a COVID-19 or suspected COVID-19 infection (still suffering or suffered symptoms) for longer than 1 week Even if your COVID-19 test result was negative, or you were not tested at all

  * Persons who are 18 years of age or older

General considerations according to Myalgic encephalomyelitis: International Consensus Criteria:

* Patients should meet the full criteria for epidemiological studies. If specific subgroups or atypical ME are included in a research study, that should be clearly indicated.
* Specificity: Because critical symptoms are compulsory, it ensures the proper selection of patients. Key operational guidelines enhance clarity and specificity. Ranking the hierarchy of the most troublesome symptoms may be helpful in some studies.
* Reliability: Symptoms must not be viewed as a nominal checklist. The International Consensus Criteria focus on symptom patterns, which increase reliability. The International Symptom Scale ensures consistency in the way questions are asked and further increases the reliability of data collected in different locations. Patients should complete the International Symptom Scale prior to entering a research study.

Exclusion Criteria:

* persons other than selected in the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People above 18 years old who have experienced covid-19 or suspected COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 2450 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Assessing and understanding acute and chronic long COVID symptoms based on a questionnaire asking different questions on testing, diagnosis, and treatments. | once through study completion, an average of one year
  List of relevant morbidities, testing, diagnosis, and treatments assessed as present/not present by medical interview (e.g. respiratory, cardiac, neurological, psychiatric diseases by interview and medical records)

SECONDARY OUTCOMES:
Assessing the long-term sequelae effects( Myalgic Encephalitis) and other comorbidities following COVID-19 vaccination. | once through study completion, an average of one year
  List of relevant symptoms or signs assessed as present/not present by medical interview (e.g. neurological impairment categories, three immune/gastro-intestinal/genitourinary impairment categories, and at least one symptom from energy metabolism/transport impairments by interview and medical records)
  The patient will meet the criteria for post-exertional neuroimmune exhaustion, at least one symptom from three neurological impairment categories, at least one symptom from three immune/gastro-intestinal/genitourinary impairment categories, and at least one symptom from energy metabolism/transport impairments according to the Myalgic Encephalitis international consensus criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
There will be no information collected that may in any way identify our patients, data will be collected via Google sheet our local collaborators will make sure all entered data is true and there is no misleading data.
  The questionnaire itself is online self administered.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Public Dataset, Open Source Code
URL: https://figshare.com/articles/dataset/Analysis_of_COVID-19_Patients_Symptoms_and_Vaccine_Impact_Using_Deep_Learning_Approach_and_Development_Machine_Learning_Based_Risk_Calculator_A_Multicentric_Collaborative_Study/25585452

REFERENCES:
- [Result] Shaheen N, Shaheen A. Long-term sequelae of COVID-19 (myalgic encephalomyelitis): An international cross-sectional study. Medicine (Baltimore). 2022 Nov 11;101(45):e31819. doi: 10.1097/MD.0000000000031819. PMID 36397426
- [Derived] Shaheen A, Shaheen N; Long COVID Collaboration Study Group in the LMICs; Shoib S, Saeed F, Buhari M, Bharmauria V, Flouty O. Deep learning analysis of long COVID and vaccine impact in low- and middle-income countries (LMICs): development of a risk calculator in a multicentric study. Front Public Health. 2025 Jun 26;13:1416273. doi: 10.3389/fpubh.2025.1416273. eCollection 2025. PMID 40642241
- See also: Deep learning analysis of long COVID and vaccine impact in low- and middle-income countries (LMICs): development of a risk calculator in a multicentric study — https://www.frontiersin.org/journals/public-health/articles/10.3389/fpubh.2025.1416273/full?fbclid=IwY2xjawKlCXlleHRuA2FlbQIxMABicmlkETFhUnlPQUpaeUFuck9rQm5VAR78-fWFJcdeLEN6QOI1a-Lbkfv80AYsLB5gsV-bjzuGWVLV9vRGUO9gzuX6ig_aem_q0WOCg_2r7hkXL-Jdjua3A
- See also: Main results paper — https://www.frontiersin.org/journals/public-health/articles/10.3389/fpubh.2025.1416273/full?fbclid=IwY2xjawKlCXlleHRuA2FlbQIxMABicmlkETFhUnlPQUpaeUFuck9rQm5VAR78-fWFJcdeLEN6QOI1a-Lbkfv80AYsLB5gsV-bjzuGWVLV9vRGUO9gzuX6ig_aem_q0WOCg_2r7hkXL-Jdjua3A
- Available data/document: Individual Participant Data Set — https://figshare.com/articles/dataset/Analysis_of_COVID-19_Patients_Symptoms_and_Vaccine_Impact_Using_Deep_Learning_Approach_and_Development_Machine_Learning_Based_Risk_Calculator_A_Multicentric_Collaborative_Study/25585452 — Open Code and Dataset

DOCUMENTS (1):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT05059184/Prot_000.pdf